CLINICAL TRIAL: NCT00605514
Title: VRC 206: A Phase I Study to Evaluate the Safety and Immunogenicity of an Ebola DNA Plasmid Vaccine, VRC-EBODNA023-00-VP, and a Marburg DNA Plasmid Vaccine, VRC-MARDNA025-00-VP, in Healthy Adults
Brief Title: Ebola and Marburg Virus Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: RCHSPB
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 080065; 08-I-0065
Record Dates: First submitted 2008-01-29; First posted 2008-01-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-06-21

CONDITIONS: Ebola Vaccines; Marburg Virus Disease; Ebola Virus Disease; Marburgvirus; Ebolavirus
Keywords: Hemorrhagic Fever; Healthy; Immunity; T-Cells; Filovirus; Healthy Volunteer; HV
MeSH Terms: conditions — Marburg Virus Disease; Hemorrhagic Fever, Ebola; Hemorrhagic Fevers, Viral

INTERVENTIONS:
Drug: VRC-EBODNA023-00-VP
Drug: VRC-MARDNA025-00-VP

SUMMARY:
This study will determine if experimental vaccines to prevent Ebola virus infection and Marburg virus infection are safe and what side effects, if any, they cause. Ebola virus infection may range from mild to severe, and may cause breathing problems, severe bleeding, kidney problems and shock that can lead to death. Marburg virus infection causes an illness similar to that caused by the Ebola virus. The vaccines used in this study contain genetic material produced in the laboratory that causes the body to make a small amount of either Ebola or Marburg virus proteins. No Ebola or Marburg virus is in the vaccines.

Normal healthy volunteers between 18 and 60 years of age may be eligible for this study.

Participants are assigned to receive injections of either the Marburg or the Ebola vaccine. The first group of participants will receive the Marburg vaccine and the second group will receive the Ebola vaccine. The injections are given at 4-week intervals (study weeks 0, 4 and 8). They are given into a muscle with a needleless system called the Biojector(Registered Trademark) 2000.

Participants keep a diary at home (on paper or electronically) for 5 days, in which they record their temperature, symptoms and any reaction at the injection site. They call a study nurse the day after vaccination to report how they feel and return to the clinic for follow-up 2 weeks after each injection (weeks 2, 6 and 10). The visits include a check of vital signs, blood and urine tests, medical history and review of medications taken. Additional visits at weeks 12, 24 and 32 include a check of vital signs, medical history and blood tests.

DETAILED DESCRIPTION:
Study Design:

This is an open label Phase I study to evaluate safety, tolerability, and immunogenicity of two recombinant DNA vaccines: one against Marburg virus infections and one against Ebola virus infections. The hypothesis is that each vaccine will be safe for human administration and elicit a humoral and T cell mediated immune response. The primary objectives are to evaluate the safety and tolerability of the investigational vaccines in healthy adults. Secondary and exploratory objectives are related to the immunogenicity of each study vaccine.

Product Description:

VRC-MARDNA025-00-VP (Marburg DNA) is composed of one closed-circular DNA plasmid encoding for the glycoprotein (GP) from the Angola strain of Marburg. VRC-EBODNA023-00-VP (Ebola DNA WT) is composed of two closed-circular DNA plasmids, one encodes for GP from the Zaire strain and one encodes for GP from the Sudan-Gulu strain of Ebola. DNA vaccine vials will be supplied at 4 mg/mL. Each DNA vaccination will be 1 mL of vaccine administered intramuscularly (IM) into the deltoid muscle using the Biojector[R] 2000 Needle-Free Injection Management System (Biojector).

Subjects:

A total of 20 healthy adults, ages 18-60 years, will be enrolled into two groups of 10 subjects each. No more than one subject per group may be in the age range of 51-60 years.

Study Plan:

Subjects will be sequentially enrolled into two groups. Group 1 subjects will receive the Marburg DNA vaccine and Group 2 subjects will receive the Ebola DNA WT vaccine. The first 3 enrollments in each group will occur no faster than one per day. Before completing enrollment into each group, there will be a study pause with review by the Protocol Safety Review Team (PSRT) when there is at least 2 weeks of safety follow-up on the third subject's first injection. Before the initiation of Group 2, the FDA must have assessed administration of the Ebola DNA WT vaccine as safe to proceed. In addition, there will be a study pause with review by the PSRT when there is at least two weeks of safety follow-up on the last subject enrolled into Group 1.

VRC 206 Group 1 will receive Marburg DNA, accrue 10 subjects and deliver injections on Day 0 with a dose 4 mg, Day 28 plus or minus 7 with a dose 4 mg and Day 56 plus or minus 7 with a dose 4 mg.

VRC 206 Group 2 will receive Ebola DNA WT, accrue 10 subjects and deliver injections on Day 0 with a dose of 4 mg, Day 28 plus or minus 7 with a dose 4 mg and Day 56 plus or minus 7 with a dose 4 mg.

The total accrual will be 20 subjects. The injections will be administered at least 21 days between DNA injections.

The original protocol design required 9 clinic visits and 3 telephone follow-up contacts for each subject.

The Version 4.0 protocol amendment allows a 4th injection for those who consent. Consent and administration of the 4th injection could occur anytime in the interval starting with Study Week 32 through Study Week 52. The 4th injection follow-up schedule includes 1 telephone contact and 4 follow-up visits after the injection.

Study Duration: The original study requires 32 weeks of clinical follow up for each participant. Subjects who consent to the amended schedule with a 4th injection will have an additional 12 weeks of follow up.

ELIGIBILITY:
* INCLUSION CRITERIA:

The following eligibility criteria apply to initial enrollment into the study:

A participant must meet all of the following criteria:

1. 18 to 60 years old
2. Available for clinical follow-up through Week 32
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
4. Complete an AoU prior to enrollment and verbalize understanding of all questions answered incorrectly
5. Able and willing to complete the informed consent process
6. Willing to donate blood for sample storage to be used for future research
7. In good general health without clinically significant medical history
8. Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) less than 40 within the 28 days prior to enrollment

   LABORATORY CRITERIA WITHIN 28 DAYS PRIOR TO ENROLLMENT:
9. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men
10. White blood cells (WBC) = 3,300-12,000 cells/mm3
11. Differential either within institutional normal range or accompanied by site physician approval
12. Total lymphocyte count greater than or equal to 800 cells/mm3
13. Platelets = 125,000 - 400,000/mm3
14. Alanine aminotransferase (ALT) less than 1.25 upper limit of normal
15. Serum creatinine less than or equal to 1 x upper limits of normal (less than or equal to1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males)
16. Normal urinalysis defined as negative glucose, negative or trace protein and no clinically significant blood in the urine
17. Negative FDA-approved HIV blood test. [Note: Results of HIV ELISA will be documented, but a negative HIV polymerase chain reaction (PCR) test result will be sufficient for eligibility screening of subjects with positive HIV ELISA that is due to prior participation in an HIV vaccine study]
18. Negative hepatitis B surface antigen (HBsAg)
19. Negative anti-HCV and negative hepatitis C virus (HCV) PCR
20. Partial thromboplastin time (PTT) within institutional normal range
21. Prothrombin time (PT) less than or equal to upper limit of normal

    FEMALE-SPECIFIC CRITERIA:
22. Negative Beta-HCG pregnancy test (urine or serum) for women presumed to be of reproductive potential
23. A female participant must meet one of the following criteria:

    * No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

OR

* Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 32 of the study,

OR

* Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 32 of the study by one of the following methods:

  1. condoms, male or female, with or without a spermicide
  2. diaphragm or cervical cap with spermicide
  3. intrauterine device
  4. contraceptive pills or patch, Norplant, Depo-Provera or any other FDA-approved contraceptive method
  5. male partner has previously undergone a vasectomy

     EXCLUSION CRITERIA:

     A SUBJECT WILL BE EXCLUDED IF ONE OR MORE OF THE FOLLOWING CONDITIONS APPLY:

     Women:
     1. Breast-feeding or planning to become pregnant during the first 32 weeks after enrollment

        SUBJECT HAS RECEIVED ANY OF THE FOLLOWING SUBSTANCES:
     2. Investigational Ebola vaccine in a prior clinical trial
     3. Immunosuppressive medications, cytotoxic medications, inhaled corticosteroids, or long-acting beta-agonists within the 12 weeks prior to enrollment. [With the exceptions that use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis, or short-acting beta-agonists in controlled asthmatics; or a short course (duration of 10 days or less, or a single injection) of corticosteroids for a non-chronic condition at least 2 weeks prior to enrollment in this study will not exclude study participation.]
     4. Blood products within 120 days prior to HIV screening
     5. Immunoglobulin within 60 days prior to HIV screening
     6. Live attenuated vaccines within 30 days prior to initial study vaccine administration
     7. Investigational research agents within 30 days prior to initial study vaccine administration
     8. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration
     9. Current anti-tuberculosis prophylaxis or therapy

        SUBJECT HAS A HISTORY OF ANY OF THE FOLLOWING CLINICALLY SIGNIFICANT CONDITIONS:
     10. Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain
     11. Idiopathic urticaria within the past 2 years
     12. Autoimmune disease or immunodeficiency
     13. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past 2 years or that requires the use of oral or parenteral corticosteroids
     14. Diabetes mellitus (type I or II), with the exception of gestational diabetes
     15. History of thyroidectomy or thyroid disease that required medication within the past 12 months
     16. A history of hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema
     17. Hypertension that is not well controlled by medication or blood pressure that is more than 145/95 at enrollment
     18. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions), significant bruising or bleeding difficulties with IM injections or blood draws, or routine use of anticoagulant medications
     19. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study
     20. Seizure disorder other than: 1) febrile seizures under the age of 2 years, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years
     21. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
     22. Allergic reaction to aminoglycoside antibiotics
     23. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide plan or attempt
     24. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a subject's ability to give informed consent

     Eligibility for the Optional 4th Study Injection:

     Eligibility to receive a 4th injection requires the original consent (Appendix I) to be reviewed again with a study clinician, as well as the consent for the optional 4th injection (Appendix V) to be reviewed and signed. To be eligible the study subject must meet the following criteria:
* Has completed the 3-injection schedule for the Group in which he/she was enrolled.
* Has remained in follow-up through Study Week 32 without any serious adverse events.
* Meets the original study eligibility criteria for hemoglobin, platelets. PT. PTT. Creatinine and ALT within the 28 days prior to the 4th injection.
* Assessed as continuing to have a healthy vaccine study volunteer status by recent interim history and appropriate physical assessments.
* If a woman of reproductive potential, is willing to continue with a pregnancy prevention method (from among those meeting the original study eligibility) through 12 weeks after the injection and is confirmed as not pregnant on the day of the 4th injection prior to administration of the injection.
* Available for clinical follow-up through 12 weeks after the 4th injection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01-25; Primary Completion 2010-06-21 (Actual); Study Completion 2010-06-21 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity, lab tests, AEs)

SECONDARY OUTCOMES:
Immunogenicity (cellular and humoral immune function assays)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Geisbert TW, Jahrling PB. Exotic emerging viral diseases: progress and challenges. Nat Med. 2004 Dec;10(12 Suppl):S110-21. doi: 10.1038/nm1142. PMID 15577929
- [Background] Meslin FX. Global aspects of emerging and potential zoonoses: a WHO perspective. Emerg Infect Dis. 1997 Apr-Jun;3(2):223-8. doi: 10.3201/eid0302.970220. PMID 9204308
- [Background] Okware SI, Omaswa FG, Zaramba S, Opio A, Lutwama JJ, Kamugisha J, Rwaguma EB, Kagwa P, Lamunu M. An outbreak of Ebola in Uganda. Trop Med Int Health. 2002 Dec;7(12):1068-75. doi: 10.1046/j.1365-3156.2002.00944.x. PMID 12460399
- [Derived] Sarwar UN, Costner P, Enama ME, Berkowitz N, Hu Z, Hendel CS, Sitar S, Plummer S, Mulangu S, Bailer RT, Koup RA, Mascola JR, Nabel GJ, Sullivan NJ, Graham BS, Ledgerwood JE; VRC 206 Study Team. Safety and immunogenicity of DNA vaccines encoding Ebolavirus and Marburgvirus wild-type glycoproteins in a phase I clinical trial. J Infect Dis. 2015 Feb 15;211(4):549-57. doi: 10.1093/infdis/jiu511. Epub 2014 Sep 14. PMID 25225676